CLINICAL TRIAL: NCT00599469
Title: Phase 1 Study to Determine the Efficacy of Using Far Infrared Radiation for the Treatment of Alzheimer's Disease.
Brief Title: Far Infrared Treatment for Alzheimer's Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: Dr. Kwasi Donyina/Founder and President, GAAD Medical Research Institute Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAAD-AD-CTP1
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2009-08-17 (Estimated); Status verified 2009-08

CONDITIONS: Alzheimer Disease
Keywords: Acute Confusional Senile Dementia; Alzheimer Type Senile Dementia; SENILE PLAQUES; NEUROFIBRILLARY TANGLES; NEUROPIL THREADS
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Far Infrared Radiation
  Interventions: Radiation: Far Infrared Radiation (5μm to 20μm wavelength)

INTERVENTIONS:
Radiation: Far Infrared Radiation (5μm to 20μm wavelength) — Far Infrared radiation for 30 to 40 minutes per treatment session.

SUMMARY:
Alzheimer's disease is a progressive and fatal brain disease. This study will investigate the use of far infrared radiation treatment for the disease.

DETAILED DESCRIPTION:
Alzheimer's destroys brain cells, causing problems with memory, thinking and behaviour severe enough to affect work, lifelong hobbies or social life. Alzheimer's gets worse over time and it is fatal.

Alzheimer's, which has no current cure, is the most common form of dementia. It is hereby postulated that far infrared radiation of the central nervous and endocrine systems will help with the management of the disease and possibly cure the disease.

ELIGIBILITY:
Inclusion Criteria:

* People with Alzheimer's disease

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-02; Primary Completion 2009-03 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Management and Cure of Alzheimer's Disease | 1 year

SECONDARY OUTCOMES:
Management and Cure of Dementia | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ken Nedd, M.D., Principal Investigator — GAAD Medical Research Institute Inc.; Kwasi Donyina, Ph.D., Study Director — GAAD Medical Research Institute Inc.
Locations (1):
- The Centre for Incurable Diseases, Toronto, Ontario, Canada